CLINICAL TRIAL: NCT04229394
Title: Phase I Safety, Tolerability, and Pharmacokinetics Study of 2ccPA in Patients With Symptomatic Knee Osteoarthritis
Brief Title: 2ccPA Study in Patients With Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OEP-2PM102-101
Record Dates: First submitted 2018-04-10; First posted 2020-01-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: 2ccPA
MeSH Terms: conditions — Osteoarthritis | interventions — 2-carba-cyclic phosphatidic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects and study site personnel (other than the study site pharmacists) are all blinded to the treatment assignment. An un-blind pharmacist is necessary for study drug preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2ccPA (Experimental): Only day 1 Intra-articular injection can be given under direct ultrasound guidance; the only one strength for 2ccPA injection vial is 2,400 μg (1.2 mL per vial).
  IP name: 2-carba-cyclic phosphatidic acid (2ccPA)
  Interventions: Drug: 2ccPA
- Placebo (Placebo Comparator): Only day 1 Intra-articular injection can be given under direct ultrasound guidance; placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 2ccPA — Four dose cohorts (50 μg, 200 μg, 800 μg, and 2,400 μg) are planned in this study sequentially.
  study group: one dose intra-articular on day1
  Other Names: 2-carba-cyclic phosphatidic acid
  Arms: 2ccPA
Drug: placebo — A total of 8 subjects will be recruited and randomized in each dose cohort with a 3:1 ratio (6 subjects in the 2ccPA treatment arm and 2 subjects in the placebo arm).
  control group: one dose intra-articular on day 1
  Arms: Placebo

SUMMARY:
This clinical trial is designed to determine safety and tolerability as well as the MTD of a single-dose 2ccPA and PK data in symptomatic knee OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative disease frequently associated with symptoms such as inflammation, stiffness, muscle weakness, joint swollen and joint pain. 2-carba-cyclic phosphatidic acid (2ccPA) is the derivative of natural occurring phospholipid mediator, cyclic phosphatidic acid (cPA). Previous studies suggested that 2ccPA inhibits inflammation and may relieve the pain caused by osteoarthritis.

This clinical study aims to assess the safety, tolerability, and pharmacokinetics as well as the maximal tolerated dose (MTD) of a single-dose 2ccPA in symptomatic knee OA. Safety and efficacy data for the design and conduction of subsequent studies will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are aged between 40 and 75 years old (inclusive)
2. Subjects diagnosed with symptomatic knee OA for at least 6 months prior to study entry (randomization)
3. Subjects whose radiographic evidence of knee OA are classified as grade II or III (according to Kellgren and Lawrence grading system)
4. Subjects with OA knee pain on the majority of days in the past 30 days prior to study entry (randomization).
5. A score of over 8 and below 16 out of 20 for the WOMAC pain subscale in the index knee in screening
6. Male subjects must agree to practice medically acceptable contraceptive regimen (i.e., sterilization surgery, barrier method, abstention) from screening visit until at least 1 month after the study treatment.
7. Subjects who are willing to sign the informed consent form (ICF)
8. Subjects with normal liver and renal function:

ALT and AST do not exceed 1.5 ULN (upper limit of normal) Serum Cr levels do not exceed 1.0 ULN

Exclusion Criteria:

1. Subjects with known hypersensitivity to study medication
2. Female subjects who are pregnant or lactating. Women of childbearing potential must agree to practice medically acceptable contraceptive regimen from screening visit until at least 1 month after the study treatment and must have a negative urine pregnancy test no earlier than 72 hours prior to study treatment.
3. Intra-articular use of corticosteroid, hyaluronic acid or other intra-articular injection in study knee within 3 months prior to study entry (randomization)
4. Use of chondroitin and/ or glucosamine within 4 weeks prior to study entry (randomization)
5. Subjects with known malignancy
6. History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, lymphoma, arthritis associated with inflammatory bowel disease, sarcoidosis and amyloidosis
7. Prior arthroscopic or open surgery on the study knee within 6 months prior to study entry (randomization)
8. Clinical signs and symptoms of active knee infection or being treated for knee infection at screening
9. Patients with active inflammation: patients with CRP higher than upper limit of normal range at screening visit will be excluded from the study.
10. Subjects with concurrent medical or arthritic condition that could interfere with evaluation of the index knee joint, including fibromyalgia, based on investigator's clinical judgment
11. More significant pain from the back or the hip than the knee
12. Skin breakdown or lesion on the study knee that is not suitable for injection, based on investigator's discretion
13. Prior knee replacement on the study knee or planned knee replacement during the study period
14. Subjects with (1) meniscus tears which requires repairment surgery OR (2) anterior cruciate ligament rupture based on screening MRI results
15. Patients with known severe synovitis, synovium necrosis in the target knee joint judged by investigator at screening
16. Patients with PT/ APTT higher than the upper limit of normal range at screening
17. History of drug or alcohol dependence in the past 3 years
18. Having known infection with HIV-1, HBV, HCV
19. Use of any investigational drug or participation in any drug study within 4 weeks prior to study entry (randomization)
20. Subjects who are unwilling or unable to comply with study procedures
21. Any clinical condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk to participate in the study or confounds the ability to interpret data from the study as judged by the investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Adverse events will be coded with MedDRA and analyzed by system organ class (SOC) and preferred term. The number of subjects who experience DLT will be calculated at each dose level and the result of MTD will be provided. | 85 days
  To determine safety and tolerability as well as the maximal tolerated dose (MTD) of a single-dose 2ccPA in symptomatic knee OA

SECONDARY OUTCOMES:
20% improvement in the The Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain and physical function subscales | 85 days
  Proportion of subjects with a 20% improvement in the WOMAC pain and physical function subscales on Day 2, Day 3, Day 8, Day 15, Day 29 post treatment, compared with placebo group and baseline
50% improvement in the The Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain and physical function subscales | 85 days
  Proportion of subjects with a 50% improvement in the WOMAC pain and physical function subscales on Day 2, Day 3, Day 8, Day 15, Day 29 post treatment, compared with placebo group and baseline
70% improvement in the The Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain and physical function subscales | 85 days
  Proportion of subjects with a 70% improvement in the WOMAC pain and physical function subscales on Day 2, Day 3, Day 8, Day 15, Day 29 post treatment, compared with placebo group and baseline
Maximum plasma concentration (Cmax) of 2ccPA | at baseline (pre-dose), 15 ± 5 minutes, 30 ± 5 minutes, 1 hour ± 10 minutes, 2 hours ± 10 minutes, 4 hours ± 10 minutes, 6 hours ± 10 minutes, 8 hours ± 10 minutes, 12 ± 2 hours, 24 ± 2 hours (Day 2) and 48 ± 2 hours (Day 3) after 2ccPA treatment.
  Pharmacokinetic profile of 2ccPA
Time to maximum plasma concentration (Tmax) of 2ccPA | at baseline (pre-dose), 15 ± 5 minutes, 30 ± 5 minutes, 1 hour ± 10 minutes, 2 hours ± 10 minutes, 4 hours ± 10 minutes, 6 hours ± 10 minutes, 8 hours ± 10 minutes, 12 ± 2 hours, 24 ± 2 hours (Day 2) and 48 ± 2 hours (Day 3) after 2ccPA treatment.
  Pharmacokinetic profile of 2ccPA
Area under plasma concentration-time curve (AUC) of 2ccPA | at baseline (pre-dose), 15 ± 5 minutes, 30 ± 5 minutes, 1 hour ± 10 minutes, 2 hours ± 10 minutes, 4 hours ± 10 minutes, 6 hours ± 10 minutes, 8 hours ± 10 minutes, 12 ± 2 hours, 24 ± 2 hours (Day 2) and 48 ± 2 hours (Day 3) after 2ccPA treatment.
  Pharmacokinetic profile of 2ccPA
Apparent total body clearance (CL/F) of 2ccPA | at baseline (pre-dose), 15 ± 5 minutes, 30 ± 5 minutes, 1 hour ± 10 minutes, 2 hours ± 10 minutes, 4 hours ± 10 minutes, 6 hours ± 10 minutes, 8 hours ± 10 minutes, 12 ± 2 hours, 24 ± 2 hours (Day 2) and 48 ± 2 hours (Day 3) after 2ccPA treatment.
  Pharmacokinetic profile of 2ccPA
Apparent volume of distribution (Vz/F) of 2ccPA | at baseline (pre-dose), 15 ± 5 minutes, 30 ± 5 minutes, 1 hour ± 10 minutes, 2 hours ± 10 minutes, 4 hours ± 10 minutes, 6 hours ± 10 minutes, 8 hours ± 10 minutes, 12 ± 2 hours, 24 ± 2 hours (Day 2) and 48 ± 2 hours (Day 3) after 2ccPA treatment.
  Pharmacokinetic profile of 2ccPA
Elimination half-life (t1/2) of 2ccPA | at baseline (pre-dose), 15 ± 5 minutes, 30 ± 5 minutes, 1 hour ± 10 minutes, 2 hours ± 10 minutes, 4 hours ± 10 minutes, 6 hours ± 10 minutes, 8 hours ± 10 minutes, 12 ± 2 hours, 24 ± 2 hours (Day 2) and 48 ± 2 hours (Day 3) after 2ccPA treatment.
  Pharmacokinetic profile of 2ccPA
Synovial fluid 2ccPA level | before intra-articular injection treatment and 24 hours ± 2 hours after intra-articular injection.
  Changes from baseline (pre-dose) in synovial fluid 2ccPA and synovial fluid matrix metalloproteinase (MMP)-1, -3 and -13 levels at 24 hours after 2ccPA treatment
Synovial fluid matrix metalloproteinase (MMP)-1 level | before intra-articular injection treatment and 24 hours ± 2 hours after intra-articular injection.
  Changes from baseline (pre-dose) in synovial fluid 2ccPA and synovial fluid matrix metalloproteinase (MMP)-1, -3 and -13 levels at 24 hours after 2ccPA treatment
Synovial fluid matrix metalloproteinase (MMP)-3 level | before intra-articular injection treatment and 24 hours ± 2 hours after intra-articular injection.
  Changes from baseline (pre-dose) in synovial fluid 2ccPA and synovial fluid matrix metalloproteinase (MMP)-1, -3 and -13 levels at 24 hours after 2ccPA treatment
Synovial fluid matrix metalloproteinase (MMP)-13 level | before intra-articular injection treatment and 24 hours ± 2 hours after intra-articular injection.
  Changes from baseline (pre-dose) in synovial fluid 2ccPA and synovial fluid matrix metalloproteinase (MMP)-1, -3 and -13 levels at 24 hours after 2ccPA treatment
Serum prostaglandin E2 (PGE2) level | at 1 hour, 12 hours, 24 hours, 48 hours, Day 8 and Day 15 (PGE2 only) after 2ccPA treatment
  Changes from baseline (pre-dose) in serum prostaglandin E2 (PGE2) levels at 30 minutes, 1 hour, 2 hours, 4 hours, 12 hours and 24 hours after 2ccPA treatment
Serum matrix metalloproteinase (MMP)-1 level | at 1 hour, 12 hours, 24 hours, 48 hours, Day 8 and Day 15 (PGE2 only) after 2ccPA treatment
  Changes from baseline (pre-dose) in serum matrix metalloproteinase (MMP)-1,at 30 minutes, 1 hour, 2 hours, 4 hours, 12 hours and 24 hours after 2ccPA treatment
Serum matrix metalloproteinase (MMP)-3 levels | at 1 hour, 12 hours, 24 hours, 48 hours, Day 8 and Day 15 (PGE2 only) after 2ccPA treatment
  Changes from baseline (pre-dose) in serum matrix metalloproteinase (MMP)-3,at 30 minutes, 1 hour, 2 hours, 4 hours, 12 hours and 24 hours after 2ccPA treatment
Serum matrix metalloproteinase (MMP)-13 level | at 1 hour, 12 hours, 24 hours, 48 hours, Day 8 and Day 15 (PGE2 only) after 2ccPA treatment
  Changes from baseline (pre-dose) in serum matrix metalloproteinase (MMP)-13,at 30 minutes, 1 hour, 2 hours, 4 hours, 12 hours and 24 hours after 2ccPA treatment
Plasma concentration of 2ccPA | at pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours and 48 hours after 2ccPA treatment
  Plasma concentration of 2ccPA at pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours and 48 hours after 2ccPA treatment
Joint space narrowing | 85 days
  To investigate joint space narrowing by MRI at Day 85, compared with baseline and the placebo group
Ectopic bone formation | 85 days
  To investigate ectopic bone formation by MRI at Day 85, compared with baseline and the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Cheng Chen, PHD, Principal Investigator — Tri-Service General Hospital
Locations (5):
- Taiwan (5):
  - Veteran General Hospital Taipei, Taipei
  - Tri-Service General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Kaohsiung Chang Gung Memorial Hospital, Taipei
  - National Cheng Kung University Hospital, Taipei